CLINICAL TRIAL: NCT07213765
Title: Short-term Antibiotic Therapy in Mycobacterium Avium Complex Pulmonary Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bin Cao (Other)
Collaborators: MicuRx (Industry); Shanghai Pulmonary Hospital, Shanghai, China (Other); Beijing Chest Hospital (Other); Anhui Chest Hospital (Other); Jiangxi Chest Hospital (Unknown); Guangzhou Chest Hospital. (Unknown)
Responsible Party: Sponsor-Investigator, Bin Cao, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-004
Record Dates: First submitted 2025-07-19; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Mycobacterium Avium Complex Pulmonary Disease
Keywords: Mycobacterium Avium Complex Pulmonary Disease; non-tuberculous mycobacterium; contezolid
MeSH Terms: interventions — contezolid; Azithromycin; Ethambutol; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contezolid shortened regimen (Experimental)
  Interventions: Drug: Contezolid; Drug: Azithromycin; Drug: Ethambutol (E); Drug: Rifampicin (R)
- Standard regimen (Active Comparator)
  Interventions: Drug: Azithromycin; Drug: Ethambutol (E); Drug: Rifampicin (R)

INTERVENTIONS:
Drug: Contezolid — contezolid 800mg po q12h*6m
  Arms: Contezolid shortened regimen
Drug: Azithromycin — azithromycin 500mg po tiw (250mg po tiw for BW under 50kg)*6m
  Arms: Contezolid shortened regimen
Drug: Azithromycin — azithromycin 500mg po tiw (250mg po tiw for BW under 50kg)*12m
  Arms: Standard regimen
Drug: Ethambutol (E) — ethambutol 25mg/kg po tiw*6m
  Arms: Contezolid shortened regimen
Drug: Ethambutol (E) — ethambutol 25mg/kg po tiw*12m
  Arms: Standard regimen
Drug: Rifampicin (R) — rifampicin 600mg po tiw (450mg po tiw for BW under 50kg)*6m
  Arms: Contezolid shortened regimen
Drug: Rifampicin (R) — rifampicin 600mg po tiw (450mg po tiw for BW under 50kg)*12m
  Arms: Standard regimen

SUMMARY:
The goal of this clinical trial is to learn if adding contezolid works to shorten the length of treatment in mycobacterium avium pulmonary disease in adults. It will also learn about the safety of extended usage of contezolid. The main questions it aims to answer are:

Does adding contezolid to standard regimen decrease the bacterial load, lesion severity and improve the life quality of patients with mycobacterium avium pulmonary disease? What medical problems do participants have when taking contezolid for an extended length? Researchers will compare standard regimen plus contezolid to standard regimen alone to see if contezolid helps further decrease the bacterial load, lesion severity and improve the life quality of patients with mycobacterium avium pulmonary disease?

Participants will:

Take contezolid and standard regimen (azithromycin, ethambutol, and rifampicin) for 6 months, contezolid is administered every day while other drugs are taken three times a week OR take standard regimen three times a week for 12 months.

Visit the clinic once every 1 month for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study and sign the Informed Consent Form.
2. Age ≥ 18 years and ≤75 years; gender unrestricted.
3. Confirmed diagnosis of MAC pulmonary disease per ATS/IDSA 2020 guidelines or Chinese Guidelines for Diagnosis and Treatment of Nontuberculous Mycobacterial Diseases (2020 edition), with imaging features consistent with nodular bronchiectatic type.
4. No prior anti-MAC treatment within the 3 months preceding screening.
5. For premenopausal women of childbearing potential who are not surgically sterile:

   Must use a medically accepted contraceptive method (e.g., intrauterine device, hormonal contraception, or condom) during the study period and for 3 months following the last dose of investigational treatment.

   Serum or urine human chorionic gonadotropin (hCG) test must be negative within 72 hours prior to enrollment.

   Must not be breastfeeding. Male patients with partners of childbearing potential must use effective contraception during the study period and for 3 months after the last dose.
6. Organ function criteria met within one week prior to enrollment:

i. Hemoglobin ≥60 g/L; ii. Neutrophil count ≥0.5 × 10⁹/L; iii. Platelet count ≥60 × 10⁹/L; iv. Serum total bilirubin ≤3 × upper limit of normal (ULN); v. Aspartate aminotransferase (AST) ≤3 × ULN; vi. Alanine aminotransferase (ALT) ≤3 × ULN; vii. Serum creatinine <2 × ULN OR creatinine clearance ≥60 mL/min; viii. Blood urea nitrogen (BUN) ≤200 mg/L; ix. Urinalysis: Proteinuria <++; if proteinuria is +, 24-hour total protein must be <500 mg.

x. Fasting blood glucose within normal range OR stable glycemic control in diabetic patients.

xi. Cardiac function: No myocardial infarction in the preceding 6 months; No unstable angina or severe arrhythmias; New York Heart Association (NYHA) functional class >II.

Exclusion Criteria:

1. History of allergy to any study drug in the treatment regimen.
2. Mixed infections with multiple mycobacteria, bacteria, fungi, or viruses (e.g., HIV coinfection).
3. Presence of congenital/acquired immunodeficiency disorders, active pulmonary malignancy (primary or metastatic), or other malignancies requiring chemotherapy/radiation therapy during the screening or study period.
4. History of solid organ transplantation.
5. Currently undergoing dialysis.
6. Uncontrolled radiation pneumonitis requiring steroid or immunoglobulin pulse therapy, active interstitial lung disease with clinical evidence, uncontrolled and significant pleural effusion or pericardial effusion.
7. Unstable systemic comorbidities including:

   Hypertensive crisis; Unstable angina; Congestive heart failure (NYHA Class III/IV); Myocardial infarction within the preceding 6 months; Severe psychiatric disorders requiring medication (e.g., schizophrenia, bipolar disorder); Severe hepatic or renal dysfunction (e.g., Child-Pugh Class C cirrhosis, eGFR <30 mL/min/1.73m²); Neurodegenerative diseases (e.g., Alzheimer's disease).
8. Poor gastrointestinal function or malabsorption syndrome.
9. Receipt of other investigational drugs within 4 weeks prior to the first study drug administration.
10. Concurrent participation in another interventional clinical trial, unless it is an observational/noninterventional study OR follow-up phase of a completed intervention trial.
11. Any physical examination findings or clinical tests deemed by the investigator as likely to:

Interfere with study results; Increase risks of complications during treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
culture conversion | end of month 6
  2 consecutive negative sputum mycobacterial culture at least 4 weeks apart, or one negative bronchoalveolar lavage fluid culture/NGS.
CT lesion absorption | end of month 6
  >30% decrease in lesion size or number of nodules measured on CT
QOL-B+NTM module | end of month 6
  Improvement greater than MID in at least 7 out of 12 domains in QOL-B with NTM-module (must include respiratory symptoms and NTM-PD symptoms)

SECONDARY OUTCOMES:
culture conversion | up to month 12
  2 consecutive negative sputum mycobacterial culture at least 4 weeks apart, or one negative bronchoalveolar lavage fluid culture/NGS.
CT lesion status | end of month 3, 6, and 12 (for standard regimen)/end of month 3 and 6 (for shortened regimen)
  >30% decrease in lesion size or number of nodules measured on CT
Questionnaire: Quality of life-bronchiectasis (QOL-B) and NTM module | up to month 12
  Improvement greater than minimal importance difference in at least 7 out of 12 domains in QOL-B with NTM module (must include respiratory symptoms and NTM-PD symptoms)
SGRQ | up to month 12
time to positivity of mycobacterium culture | up to month 12

OTHER OUTCOMES:
Number of participants with adverse events | up to month 12
  Adverse events related to study intervention (short-term regimen and standard regimen) are reported by participants.
MAC strain drug-sensitivity | end of month 6 (for shortened regimen)/end of month 12 (for standard regimen)
  Phenotypic drug sensitivity will be evaluated with microdilution method for macrolides, amikacin, rifampicin, and ethanmbutol
Number of participants with treatment-related abnormal laboratory tests results | up to month 12
  Laboratory tests include complete blood count, liver function and kidney function. Abnormalities will be recorded and discussed to determine the causality between treatment and laboratory findings.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojin Cui, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (6):
- China (6):
  - Anhui Chest Hospital, Hefei, Anhui
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Guangzhou Chest Hospital, Guangzhou, Guangdong
  - Jiangxi Chest Hospital, Nanchang, Jiangxi
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No